CLINICAL TRIAL: NCT04346810
Title: Burnout Among Caregivers Facing COVID-19 Health Crisis at a Non-conventional Intensive Care Unit Compared to a Conventional Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Raymond Poincaré (Other)
Collaborators: Dominique FLETCHER MD-PhD (Unknown); Guillaume GERI MD-PhD (Unknown); Clement DURET MD (Unknown)
Responsible Party: Principal Investigator, HARKOUK Hakim, Principal Investigator, Hôpital Raymond Poincaré
Other Study IDs: CSC19APR
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Burnout, Caregiver; Intensive Care Unit; Stress, Psychological
MeSH Terms: conditions — COVID-19; Caregiver Burden; Stress, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recovery room caregivers: Caregivers working at a recovery room shifted into an intensive care unit for the management of patients suffering from coronavirus infection and needing a resuscitation
  Interventions: Other: Patient management suffering of coronavirus infection
- Intensive care unit caregivers: Caregivers working at a conventional intensive care unit for the management of patients suffering from coronavirus infection and needing a resuscitation
  Interventions: Other: Patient management suffering of coronavirus infection

INTERVENTIONS:
Other: Patient management suffering of coronavirus infection — Welle-being and stress of the caregivers

SUMMARY:
The intense health crisis due to COVID-19 led to a profound reorganization of the activities at theatres, recovery rooms and the intensive care units. The caregivers are facing several issues and are daily exposed to an intensification of the work. Assessing the stress and the well-being of the caregivers is very important in this context.

DETAILED DESCRIPTION:
The current period of intense and prolonged health crisis has necessitated a profound reorganization of the activities and organizations of the intensive care hospital services in order to be able to cope with it.

Caregivers are at the heart of the management of this crisis and are exposed daily to these situations of repeated emergencies, an intensification of the pace of work and difficulties in care.

In this context, it seemed important to us to try to quantify this pressure of care, in order to be able to offer in second care adapted to caregivers who would like it.

The assessment of the mental state of the caregivers as well as the collection of the feelings and perceptions on the current crisis and its management will be carried out by anonymous and voluntary self-questionnaire in collaboration with the service of professional pathologies and occupational medicine of the hospital structure

ELIGIBILITY:
Inclusion Criteria:

* Consent to participation; caregivers working at recovery room; caregiver working at intensive care unit

Exclusion Criteria:

* refusal of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers working in the recovery room shifted into an intensive care unit or in the conventional intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Stress in a recovery room transformed into an intensive care unit versus a conventional intensive care unit | A 3 months period from the starting of the pandemic
  stress level of caregivers managing patients with coronavirus infection needing airway support or resuscitation. The level of stress will be quantified with the Maslach burnout Inventory.

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers

REFERENCES:
- [Background] Staloff J, Diop M, Matuk R, Riese A, White J. Caring for Caregivers: Burnout and Resources for Caregivers in Rhode Island. R I Med J (2013). 2018 Nov 1;101(9):10-11. No abstract available. PMID 30384512
- [Background] Pastores SM. Burnout Syndrome in ICU Caregivers: Time to Extinguish! Chest. 2016 Jul;150(1):1-2. doi: 10.1016/j.chest.2016.03.024. No abstract available. PMID 27396768